CLINICAL TRIAL: NCT06536374
Title: A Phase II, Open Label, Randomized Controlled Pilot Study Evaluating Trimethoprim in Patients Commencing Androgen Deprivation Therapy for Prostate Cancer
Brief Title: Folate Study in Men With Advanced Prostate Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Michael Liss, Associate Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 812072
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer
Keywords: Androgen deprivation therapy; Folic Acid
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Trimethoprim

STUDY DESIGN:
Intervention Model Description: This study is a Phase II, open label, randomized controlled trial. Subjects will be randomized 1:1 to either Trimethoprim (TMP) + androgen deprivation therapy per standard of care or to androgen deprivation therapy alone.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Trimethoprim plus androgen deprivation therapy (Experimental): Administration of trimethoprim to reduce folic acid levels at the time of standard of care androgen deprivation therapy.
  Interventions: Drug: Trimethoprim Tablets
- Standard of Care treatment (No Intervention): Standard of care treatment participants will have no intervention, only their prescribed androgen deprivation therapy.

INTERVENTIONS:
Drug: Trimethoprim Tablets — Trimethoprim 150mg is administered once daily for 3 months
  Arms: Trimethoprim plus androgen deprivation therapy

SUMMARY:
The researchers hope to learn if Trimethoprim, 150mg taken daily for 3 months, is a safe and effective way to reduce folate levels at time of Androgen Deprivation Therapy (ADT) in men with advanced prostate cancer.

This study will help find out what effects, good and/or bad, this drug has on people who take it and on its effect on the disease. The safety of this drug in humans has been tested in prior research studies; however, some side effects may not yet be known.

DETAILED DESCRIPTION:
While taking part in this study, participants will be asked to attend approximately 4 to 7 visits - depending on what randomized arm they are in - with the researchers or study staff.

It may be necessary for participants to return to the hospital/clinic every 1-3 months as part of their regular care. Research procedures will be completed at the same time as these routine standard of care visits. Participants will be asked to stop taking any supplements or medications containing folic acid or potassium prior to enrolling in the study.

ELIGIBILITY:
INCLUSION CRITERIA

1. Provision of signed and dated informed consent form.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Age ≥ 18 years.
4. Proven diagnosis of prostate cancer (intermediate unfavorable risk, high risk, very high risk localized per the 2025 NCCN guidelines), or metastatic hormone-sensitive prostate cancer with confirmation by pathology report and most recent prostate biopsy procedure note.
5. Prostate cancer treatment naïve.
6. Commencing androgen deprivation therapy for prostate cancer within 4 weeks of enrollment in the study. Note that radiotherapy and androgen receptor pathway inhibitors, apart from abiraterone, are allowed in both arms.
7. Hemoglobin ≥ 11 g/dL.
8. Red blood cell folate > 750 nmol/L.
9. Homocysteine < 15 micromol/L.
10. Creatine clearance within the normal range.
11. Eastern Cooperative Oncology Group performance status 0-1
12. Stated willingness to abstain from consumption of any supplements or medications containing folic acid or potassium.
13. Ability to take oral medications and be willing to adhere to trimethoprim and androgen deprivation therapy regimens.
14. For participants able to cause a pregnancy: use of condoms or other methods to ensure effective contraception with partner.
15. Agreement to adhere to lifestyle considerations described in the protocol throughout study duration.

EXCLUSION CRITERIA

1. Current use of memantine, phenytoin, and any medications that may significantly interact with TMP, including prohibited concomitant medications listed in the protocol.
2. Current use of medications that would interfere with folate metabolism (for example, methotrexate).
3. Treatment with another investigational drug while on this study.
4. Treatment with hormone therapy, immunotherapy, chemotherapy and/or radiation therapy for any malignancies within the past 2 years. Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
5. History of renal or hepatic disease, including history of hepatitis B and C.
6. Recurrent urinary tract infections, urinary retention, or neurological conditions affecting bladder function.
7. Known hypersensitivity or allergy to trimethoprim.
8. Hematological disorders (including megaloblastic anemia).
9. Commencing chemotherapy for metastatic prostate cancer.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Safety of Trimethoprim | From first dose of study therapy through 1 month after completion of study therapy.
  Proportion of participants with adverse events and serious adverse events as graded by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE).

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Liss, MD, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No